CLINICAL TRIAL: NCT06289946
Title: Topical Nitroglycerin Prior to Trans-radial Coronary Angiography: a Phase 2, Randomized Controlled Trial
Brief Title: Topical Nitro or Placebo Pre-Cath
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NitroRadialLHC
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo arm (Placebo Comparator): Subject will get placebo
  Interventions: Drug: Placebo
- Nitro arm (Experimental): Subject will get Nitrobid
  Interventions: Drug: NitroBid

INTERVENTIONS:
Drug: NitroBid — We will apply nirobid to the wrist prior to left heart catheterization.
  Arms: Nitro arm
Drug: Placebo — We will apply placebo moisturizing cream to the wrist
  Arms: Placebo arm

SUMMARY:
Phase 2, single-center, randomized, blinded clinical study to assess the safety and efficacy of topical nitroglycerin on ease of TRA during scheduled PCI. We will compare topical nitroglycerin to placebo applied prior to planned, non-urgent PCI to determine if nitroglycerin is associated with decreased number of arterial puncture attempts made, decreased time to radial access, and lower crossover rate to TFA. Subjects will be randomized to receive either topical nitroglycerin ointment or placebo prior to scheduled PCI. There will be 256 subjects enrolled in this study with 1:1 randomization.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) procedures performed by entering the radial artery, or the transradial approach (TRA), is associated with reduced vascular access site complications, bleeding, and length of hospital stay, as well as greater patient satisfaction when compared to the transfemoral approach. One of the major challenges to a successful TRA remains the small size of the radial artery. The potential need for larger catheters during PCI has been one factor limiting broader adoption of TRA and a common reason for crossover from TRA to femoral access intraprocedurally. Additionally, multiple unsuccessful attempts to access the radial artery leads to unnecessary bleeding and may lead to severe arterial vasospasms. Nitroglycerin, a vasodilator, is available in a topical form and may be used prior to PCI to dilate the radial artery and potentially increase the rate of successful TRA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female > 18 years of age at the time of consent
2. Scheduled to undergo PCI using TRA in the cardiac catheterization laboratory
3. Able to provide informed consent with capacity, given in English.

Exclusion Criteria

Patients with any of the following characteristics or conditions will not be included in the study:

1. Known nitrate allergy
2. Allergy to CeraVe Moisturizing lotion
3. Baseline hypotension with systolic blood pressure <90mmHg
4. Absence of radial artery blood flow in one or both arms
5. Presence or history of liver, rheumatologic, or chronic kidney disease
6. Current treatment with any vasodilator therapy (eg. Sildenafil)
7. Radial artery catheterization <30 days prior to enrollment
8. Active site infection
9. AV-fistula or prior radial artery harvest for bypass surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Crossover rate | 1 year
  • Evaluate number of attempts needed prior to successful radial artery cannulation and need for conversion to transfemoral approach

IPD SHARING:
Plan to Share IPD: Undecided